CLINICAL TRIAL: NCT06323278
Title: Evaluation of the Cognitive Stimulation Treatment in Patients With Parkinson's Disease
Brief Title: Effectiveness of Cognitive Stimulation Treatment in Patients With Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: PD&REHAB
Record Dates: First submitted 2024-03-06; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; GBA gene mutation; Cognitive training; Psychological and behavioral aspects
MeSH Terms: conditions — Parkinson Disease | interventions — Cognitive Training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD with GBA gene mutation: Patients with Parkinson's disease and GBA gene mutation treated with cognitive training
  Interventions: Behavioral: Cognitive training
- PD without genetic mutation: Patients with Parkinson's disease without genetic mutation treated with cognitive training
  Interventions: Behavioral: Cognitive training

INTERVENTIONS:
Behavioral: Cognitive training — The training, provided by normal clinical practice, will consist of two cycles of cognitive stimulation (8 sessions each) structured and aimed at maintaining and learning compensatory strategies that take advantage of the integrated cognitive skills.

SUMMARY:
The goal of this observational study is to evaluate the relationship between GBA mutation and cognitive stimulation treatment response in patients with Parkinson's disease. The main questions it aim to answer are: • assess whether the GBA mutation is associated with greater or lesser response to cognitive training treatment compared to a control group of PD patients without genetic mutations. • investigate the effect of cognitive stimulation program on behavioural aspects as secondary consequence induced by the possible improvement of cognitive abilities following treatment.

Participants will be undergo to: - a neuropsychological evaluation describing their cognitive profile; - a genetic investigation and finally included in a cognitive stimulation programs according to regular clinical practice. Researchers will compare PD patients with GBA mutation and patients without genetic mutation to evaluate the effectiveness of cognitive stimulation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease according to the Gelb et al. criteria;
* Patients who have carried out genetic screening for MP;
* Patients who have a raw score in the range 15.50 to 22.23 at Montreal cognitive assessment (MoCA);
* Patients who have signed the informed consent and the Privacy Policy;
* Patients who are included in cognitive stimulation programs according to regular clinical practice.

Exclusion Criteria:

* Patients with the initial suspicion of MP that during the diagnostic work-up they were suffering from a different pathology;
* Patients who have refused consent to participate in the study;
* Patients with a diagnosis of MP and cognitive profile of dementia;
* Patients undergoing deep brain neurostimulation (DBS-STN) treatment. Patients treated with DBS-STN were excluded because such treatment involves a surgical procedure whose effects on cognitive functioning could represent an interfering variable.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Experimental group: 34 PD patients with GBA gene mutation and undergoing cognitive stimulation treatment;
  * Control group: 34 patients with idiopathic PD without known genetic mutation undergoing cognitive stimulation treatment.
  The allocation of subjects to the two groups will be paired (1:1) by age ( 2 aa), sex, staging and duration of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the cognitive training on cognitive function in PD patients with GBA mutation compared to a control group of PD patients without genetic mutations. | Baseline and Six months follow-up post cognitive training
  Improvement in cognitive function after eight weeks of cognitive training as measured by the battery of italian neuropsychological tests (pencil/computer paper). The neuropsychological battery consists of domain-specific cognitive tests that will provide an aggregate measure of cognitive improvement between pre and post-treatment. Higher score indicates an improvement on cognitive function.

SECONDARY OUTCOMES:
The effect of cognitive training on behavioural aspects in PD patients. | Baseline and Six months follow-up post cognitive training
  Cognitive Reserve (CR) is a concept based on the plasticity of the brain and an higher CR lowers the risk for incidence of dementia. The CRIq consists of 20 questions collecting demographic information, the number of years of education, and occupational and leisure activities throughout adulthood including the frequency of the activities.
The effect of cognitive training on behavioural aspects in PD patients. | Baseline and Six months follow-up post cognitive training
  Beck Depression Inventory 2 (BDI-II): is a 21-item self-administered inventory designed to measure the intensity of depressive symptoms. Items are rated on a 4 point scale, with total scores obtained by summing the ratings for all items. Scores ranging between 0 and 13 are indicative of minimal depression. Scores ranging between 14 and 19 are indicative of mild level of depression while a score rangin from 29 to 63 is labeled severe.
The effect of cognitive training on behavioural aspects in PD patients. | Baseline and Six months follow-up post cognitive training
  Self-Rating Anxiety Sate (SAS): The SAS is a 20-item self-report assessment device built to measure anxiety levels, based on scoring in 4 groups of manifestations: cognitive, autonomic, motor and central nervous system symptoms. Each question is scored on a Likert-type scale of 1-4 (based on these replies: "a little of the time", "some of the time", "good part of the time", "most of the time"). The total raw scores range from 20 to 80. Higher score indicates higher anxiety levels.
The effect of cognitive training on behavioural aspects in PD patients. | Baseline and Six months follow-up post cognitive training
  Instrumental Activities of Daily Living (IADL): Instrumental activities of daily living (IADLs) are those activities that allow an individual to live independently in a community and can significantly improve the quality of life. The final total score ranges from 0 (low function, dependent) to 8 (high function, independent).
The effect of cognitive training on behavioural aspects in PD patients. | Baseline and Six months follow-up post cognitive training
  Instrumental Activities of Daily Living (IADL): Instrumental activities of daily living (IADLs) are those activities that allow an individual to live independently in a community and can significantly improve the quality of life. The final total score ranges from 0 (low function, dependent) to 8 (high function, independent).the higher the score, the greater the person's abilities.
The effect of cognitive training on behavioural aspects in PD patients. | Baseline and Six months follow-up post cognitive training
  IActivities of daily living (ADL): the ADL refers to activities oriented toward taking care of one's own body. These activities are fundamental to living in a social world; they enable basic survival and well-being, such as bathing, toileting, dressing and eating. Total score: between 6 (maximum performance) and 0 (lack of performance). the higher the score, the greater the person's abilities.
The effect of cognitive training on behavioural aspects in PD patients. | Baseline and Six months follow-up post cognitive training
  Visual Analog Scale (VAS) on the degree of expectation and subsequently on the degree of benefit of treatment, ranges from 0 (low benefit) to 10 (high benefit).
The effect of cognitive training on behavioural aspects in PD patients. | Baseline and Six months follow-up post cognitive training
  Parkinson's Disease Quality of Life 8 Questions (PDQ-8). The PDQ-8 is a self-administered questionnaire, used to measure quality of life in persons with Parkinson's disease. Each question is scored from 0-4 points and the scores are summed. The summed score is then divided by total possible score and given as a percentage score out of 100. A higher score represents a worse quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy